CLINICAL TRIAL: NCT03585075
Title: Caractérisation de l'Autofluorescence Des Tissus Sains et Pathologiques Des Cordes Vocales
Brief Title: Characterization of the Autofluorescence of Healthy and Pathological Tissues of Vocal Cords
Acronym: FLUOROCORD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2014/216
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Laryngeal Neoplasms
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this clinical trial is to provide information about autofluorescence of pathological versus healthy vocal folds tissues.

Experimentations are performed on vocal folds biopsies obtained from patients, surgered at ENT department, university hospital of Besançon. After being extracted, samples of vocal folds are submitted to excitations at 365 nm, 405 nm and 450 nm; light spectral absorptions are measured, and results are compared to reference anatomopathology.

ELIGIBILITY:
Inclusion Criteria:

* patient view in ENT department, presenting vocal fold lesion that necessitate biopsy
* patient informed and with non opposition

Exclusion Criteria:

* small (<1mm) and/or brittle sample
* Patients in emergency situations, pregnant or nursing mothers, persons deprived of their liberty, minors or protected adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples of vocal folds from ENT surgery department, University Hospital of Besançon
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
hyperspectral fluorescence of vocal folds | 30 minutes after biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No